CLINICAL TRIAL: NCT05441761
Title: Phase I/II Clinical Study of Mitoxantrone Hydrochloride Liposomes in Combination With Gemcitabine, Dexamethasone, and Cisplatin in Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: Mitoxantrone Hydrochloride Liposomes in Combination With GDP in Relapsed/Refractory PTCL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-014
Record Dates: First submitted 2022-06-23; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Treatment; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Gemcitabine; Dexamethasone; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- liposomal mitoxantrone hydrochloride (Experimental): Patients with recurrent and refractory peripheral T-cell lymphoma will receive sequentially higher doses of liposomal mitoxantrone hydrochloride in combination with gemcitabine, dexamethasone, and cisplatin for 6 cycles (planned) (21 days per cycle).
  Interventions: Drug: liposomal mitoxantrone hydrochloride, gemcitabine, dexamethasone, and cisplatin

INTERVENTIONS:
Drug: liposomal mitoxantrone hydrochloride, gemcitabine, dexamethasone, and cisplatin — Drug: Liposomal mitoxantrone hydrochloride (12 mg/m2, 16 mg/m2, 20 mg/m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Drug: gemcitabine (1000 mg/m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.
  Drug: dexamethasone (40 mg) will be administered on day 1-4 of each 21-day cycle.
  Drug: cisplatin (75 mg/m2) will be administered by an intravenous infusion on day 1 of each 21-day cycle.

SUMMARY:
This is a prospective, open-label, single arm, multicenter clinical study to evaluate the safety, tolerability, efficacy mitoxantrone hydrochloride liposome in combination with gemcitabine, dexamethasone, and cisplatin in relapsed/refractory peripheral T-cell lymphoma

DETAILED DESCRIPTION:
This is a prospective, open-label, single arm, multicenter clinical study to explore the maximum tolerated dose (MTD) of liposomal mitoxantrone hydrochloride when combined with gemcitabine, dexamethasone, and cisplatin in patients with relapsed or refractory peripheral T-cell lymphoma. Liposomal mitoxantrone hydrochloride will be given on day 1 at three different doses (12 mg/m2，16 mg/m2, 20 mg/m2) and be combined with gemcitabine, dexamethasone, and cisplatin. The dose limited toxicity (DLT) will be evaluated after the first cycle of therapy. A maximum of 6 cycles of therapy are planned. An dose expansion study of mitoxantrone hydrochloride liposome at RP2D dose level combined with gemcitabine, dexamethasone, and cisplatin was conducted to explore the efficacy and safety tolerance of the combined regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent
2. Age ≥18, ≤75 years, no gender limitation
3. Expected survival ≥ 3 months;
4. Histologically confirmed diagnosis of peripheral T-cell lymphoma, is one of the following subtypes (1) Peripheral T-cell lymphoma non-specific type (PTCL-NOS) (2) Angioimmunoblastic T-cell lymphoma (AITL) (3) Anaplastic large cell lymphoma (ALCL), ALK+ (4) Anaplastic large cell lymphoma (ALCL), ALK- (5) Other subtypes of PTCL that the researcher considered to be included in the group;
5. The criteria for relapsed/refractory lymphoma: Relapsed lymphoma is defined as lymphoma that relapsed after a complete response (CR) was achieved with initial chemotherapy. Refractory lymphoma is diagnosed by meeting any of the following criteria: 1) tumor reduction < 50% or disease progression after 4 cycles of standard regimens of chemotherapy; 2) CR was achieved by standard chemotherapy, but relapse occurred within six months; 3) Two or more times of recurrence after CR; 4) Relapse after hematopoietic stem cell transplantation;
6. There must be at least one evaluable or measurable lesion meeting lugano2014 criteria: for lymph node lesions, the length and diameter should be > 1.5cm; For non lymph node lesions, the length and diameter should be > 1.0cm;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2；
8. Bone marrow function: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelet count (PLT) ≥75×109/L, Hemoglobin(HB)≥ 80g/L(Bone marrow invasive patient ANC≥1.0×109/L,PLT≥50×109/L,HB≥75 g/L)
9. Liver and kidney function：Total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN) , The liver invasion≤3.0×ULN）;Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN , The liver invasion≤5.0×ULN; Serum creatinine (Scr) ≤1.5× ULN

Exclusion Criteria:

1. The subject had previously received any of the following anti-tumor treatments:

   1. Those who have previously received mitoxantrone or mitoxantrone liposomes;
   2. Previously received doxorubicin or other anthracycline treatment, and the total cumulative dose of doxorubicin is more than 550 mg/m2 (1 mg doxorubicin converted from other anthracycline drugs is equivalent to 2 mg epirubicin);
   3. Have received anti-tumor treatment (including chemotherapy, targeted therapy, hormone therapy, taking traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received clinical trial drugs within 4 weeks before the first use of the study drugs;
   4. Patients who have received autologous hematopoietic stem cell transplantation or allogeneic hematopoietic stem cell transplantation within 100 days of the first medication;
2. Hypersensitivity to any study drug or its components;
3. Non controlled systemic diseases (such as active infection, non controlled hypertension, diabetes, etc.)
4. Heart function and disease meet one of the following conditions:

   1. Long QT c syndrome or QTc interval > 480 ms;
   2. Complete left bundle branch block, grade II or III atrioventricular block;
   3. Serious and uncontrolled arrhythmias requiring drug treatment;
   4. New York Heart Association grade ≥ III;
   5. Cardiac ejection fraction (LVEF)< 50%;
   6. A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.
   7. Baseline NT-proBNP is greater than 800pg/ mL, cTnI is greater than the normal upper limit of our center, and the retest in three days which is still higher than the above range.
5. Hepatitis B, Hepatitis C infection in active stage (if there is a positive hepatitis B surface antigen or core antibody, additional test HBV DNA, Hepatitis B virus DNA more than 1x103 copies /mL excluded; If HCV anti-body is positive, add test for HCV RNA, and exclude HCV RNA over 1x103 copies /mL)
6. Past or current co-occurrence of other malignancies (except effectively controlled non-melanoma cutaneous basal cell carcinoma, breast/cervical carcinoma in situ, and other malignancies effectively controlled without treatment within the past five years)
7. Have primary or secondary central nervous system (CNS) lymphoma or a history of CNS lymphoma at the time of recruitment;
8. Pregnant and lactating women and patients of childbearing age who do not want to use contraception;
9. Conditions that other researchers deem inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose（RP2D） | 1 year
  To identify the RP2D
Objective response rate (ORR) | 3 year
  The ORR was defined as the proportion of patients who achieved CR or PR

SECONDARY OUTCOMES:
Dose limited toxicities (DLTs) | 1 year
maximum-tolerated dose(MTD) | 1 year
The incidence of AE and SAE | 3 year
Complete response rate (CRR) | 3 year
Duration of Response（DOR） | 3 year
progression-free survival（PFS） | 3 year
Overall survival（OS) | 3 year

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Hospital, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No